CLINICAL TRIAL: NCT04776460
Title: The Distribution of Body Constitutions Among Hong Kong Elderly Population: A Cross-sectional Study
Status: Completed | Type: Observational
Sponsor: Hong Kong Baptist University (Other)
Collaborators: The Hong Kong Jockey Club Charities Trust (Other)
Responsible Party: Principal Investigator, ZhaoXiang Bian, Chair Professor, Hong Kong Baptist University
Other Study IDs: HKBU JC 004
Record Dates: First submitted 2020-07-26; First posted 2021-03-01 (Actual); Last update posted 2021-03-01 (Actual); Status verified 2021-02

CONDITIONS: Nine Body Constitutions

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional

SUMMARY:
Hong Kong, similar as other developed economic entities, has been faced big challenges from increasing medical burden and aged population. Based on the updated estimates of domestic health expenditure by Food and Health Bureau HKSAR, the total health expenditure amounted to HK$112,144 million in 2012/13 with increasing approximate 4 times than 1992/93. According to the data from Census and Statistics Department, in 2010, there was still 13% population aged above 65 years, while in 2039, this percentage will be elevated to 28% (http://www.censtatd.gov.hk/hkstat/sub/so20.jsp). In other words, every three individuals will contain a person aged above 65 years in the future 30 years. Therefore, how to release the medical burden resulted from aged tendency of population is the critical question in optimizing the treatment expenses.

Our aims in the cross-sectional study are to 1) estimate the number and percentage of nine body constitutions among population aged 65 and over in Hong Kong 2) identify the associations between nine body constitutions and other predetermined factors such as gender, weight, diet, body mass index (BMI), blood pressure, quality of life scale scores, et al.

ELIGIBILITY:
Inclusion Criteria:

* aged 65 and over
* capable of consenting and have agreed to participate, ambulatory, and not receiving treatment modalities, which, if omitted, may result in immediate life threatening risk such as chemotherapy or radiotherapy for cancer, or dialysis for renal failure

Exclusion Criteria:

* neurological disorders such as dementia

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Study Population: The study will select the populations of aged 65 and over as subjects. We aims to cover 0.5% of these population and then 5,300 participants will be recruited from public. The random core sample will be obtained using stratified random sampling, where residential address will be randomly sampled in all 18 districts in Hong Kong with sample size proportionate to each of the district populations. We will invite them to enroll in our Chinese medicine preventive study and consent form will also be sent by mail, email and Whatsapp Business.
Sampling Method: Probability Sample
Enrollment: 5300 (Actual)
Dates: Start 2020-04-29 (Actual); Primary Completion 2021-02-03 (Actual); Study Completion 2021-02-03 (Actual)

PRIMARY OUTCOMES:
Distribution of nine body constitutions assessed by the TCM Body Constitution Questionnaire (For Elderly People) (Cantonese version) | through study completion, an average of 1 year
  The primary outcome will be the distribution of nine body constitutions in Hong Kong aged 65 and over population.

SECONDARY OUTCOMES:
Correlation between body constitution distribution and other predetermined factors | through study completion, an average of 1 year
  Secondary outcomes will be the correlation between body constitution distribution and other predetermined factors such as gender, age, weight, dietary habit, education and quality of life scores (SF-36 Hong Kong questionnaire), et al.

CONTACTS AND LOCATIONS:
Overall Officials: Zhao-xiang Bian, PhD, Principal Investigator — Hong Kong Baptist University
Locations (1):
- School of Chinese Medicine, Hong Kong Baptist University, Hong Kong, Hong Kong, China